CLINICAL TRIAL: NCT00082121
Title: Safety and Efficacy of TP10, a Complement Inhibitor, in Adult Women Undergoing Cardiopulmonary Bypass Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avant Immunotherapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: TP10-ACS-002
Record Dates: First submitted 2004-04-29; First posted 2004-05-04 (Estimated); Last update posted 2007-07-20 (Estimated); Status verified 2007-07

CONDITIONS: Myocardial Ischemia; Coronary Arteriosclerosis; Aortic Valve Insufficiency; Mitral Valve Insufficiency
Keywords: cardiac bypass; CABG; complement activation
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease; Aortic Valve Insufficiency; Mitral Valve Insufficiency

INTERVENTIONS:
Drug: TP10

SUMMARY:
The purpose of this study is to determine if the study drug (TP10), which blocks complement release, can reduce such side effects of complement inflammation as chest pain or heart attacks and be taken safely in women who undergo cardiopulmonary bypass surgery.

DETAILED DESCRIPTION:
During cardiac surgery, a substance called "complement" is released by the body. This complement causes inflammation, which can lead to side effects such as chest pain, heart attacks, or heart failure. The purpose of this study is to determine if the study drug (TP10), which blocks complement release, can reduce such side events and be taken safely in women.

ELIGIBILITY:
Inclusion Criteria:

* Female
* To undergo high-risk cardiac surgery with cardiopulmonary bypass pump (CPB)
* CABG alone or with valve surgery

Exclusion Criteria:

* Acute myocardial infarction (heart attack) within a 3 days of entering the study
* Conditions that may interfere with interpretation of electrocardiogram data
* History of immune deficiency syndrome
* Planned supplemental cardiac surgery or other surgery
* Pregnancy or lactation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-04; Study Completion 2005-12

PRIMARY OUTCOMES:
Reduction in death & myocardial infarction (MI)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - San Francisco, California
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Orlando, Florida
  - Sarasota, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Towson, Maryland
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Detroit, Michigan
  - Lansing, Michigan
  - Cincinnati, Ohio
  - Memphis, Tennessee
  - Houston, Texas
  - Danville, Virginia
  - Madison, Wisconsin
  - Milwaukee, Wisconsin